CLINICAL TRIAL: NCT07206641
Title: The Effect of Inspiratory Exercises on Diaphragm and Intercostal Muscle Thickness in Stroke Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MarmaraU-FTR-OK-1
Record Dates: First submitted 2025-09-04; First posted 2025-10-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Stroke; IMT; Inspiratory Muscle Training; Diapragm Thickness; Intercostal muscle thickness
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GROUP 1: Patients diagnosed with stroke who will be followed with inspiratory strengthening exercise

SUMMARY:
The aim of this study is to investigate the effect of inspiratory muscle strengthening exercises on bilateral parasternal intercostal muscle thickness and bilateral diaphragm muscle thickness in stroke patients and to present new data on whether the possible effect on the affected side can be associated with changes in respiratory parameters. Furthermore, as previous literature has shown that 4-week exercise programs are more effective than >6-week exercise programs, an interim assessment is planned for the second week of treatment in this study to evaluate shorter-term changes. Four weeks after completion of the exercise program (in the 8th week), patients will be re-evaluated to track potential short-term effects.

DETAILED DESCRIPTION:
Respiratory muscles consist of three main groups that control ventilation: primary inspiratory muscles, secondary inspiratory muscles, and expiratory muscles. The primary inspiratory muscle is the diaphragm, a thin dome-shaped muscle located between the thorax and the abdomen. The diaphragm, the most important respiratory muscle, contributes to 60-80% of the ventilation needs of the human body. However, the diaphragm is not the only inspiratory muscle involved in ventilation. When the load on the diaphragm increases, accessory inspiratory muscles such as the parasternal intercostal muscles, external intercostal muscles, scalene muscles, and sternocleidomastoid muscles are recruited to assist inspiration.

Involvement of the diaphragm and other respiratory muscle groups is a common condition after stroke. Due to the loss of central motor control in stroke patients, contralateral diaphragmatic weakness is observed. The thickness of the diaphragm affected by stroke is approximately 50% of that of age- and sex-matched healthy adults, as shown in studies.

After stroke, the decrease in respiratory muscle strength on the hemiplegic side may lead to pulmonary ventilation and diffusion dysfunction, reduced coughing ability, increased incidence of pulmonary complications, and reduced cardiopulmonary endurance and trunk balance control. Respiratory muscle strengthening exercises are used as an effective method in reducing these problems.

Patients diagnosed with stroke who will be followed with inspiratory strengthening exercises will be monitored by comparing the muscle thicknesses of the affected side and the healthy side. After receiving training on inspiratory strengthening exercises to be given to them, patients will regularly perform these exercises at home, and the consistent correct performance of these exercises will be monitored by a researcher through video calls with the participants over the internet.

Intercostal Muscle Thickness Measurement:

Stroke can affect the functions of respiratory muscles, particularly the accessory respiratory muscles (including the intercostal muscles), due to central nervous system damage. This condition may lead to disturbances in the breathing pattern and hypoxia.

Ultrasonography is used as an easily accessible, inexpensive, and rapid assessment method. It allows visualization of muscle contractions and has been shown to reliably evaluate both diaphragm thickness and intercostal muscle thickness. In this study, ultrasonography will be used to examine the structure and function of the intercostal muscles and to measure muscle thickness at the end of inspiration and expiration.

All patients will be placed in the supine position, and as previously demonstrated by De Troyer, A. et al., data will be obtained from the 2nd intercostal space-which is the most stable and distinct space for evaluating parasternal intercostal muscles-2 to 4 cm lateral to the sternum. After an optimal 2D image is obtained, the intercostal muscle will be evaluated and measured at end-inspiration and end-expiration. A high-frequency linear probe of 6-13 MHz, placed vertically on the chest wall with minimal pressure, will be used.

Intercostal muscle contractility can be evaluated by changes in muscle thickness (the intercostal thickness fraction (ICTf) measured using ultrasonography).

ICTf = (end-inspiration intercostal muscle thickness - end-expiration intercostal muscle thickness) / end-expiration intercostal muscle thickness × 100%

Diaphragm Muscle Thickness Measurement:

After stroke, the diaphragm, one of the primary inspiratory muscles, is prone to atrophy due to central nervous system disorders. Atrophy of the diaphragm leads to decreased exercise capacity associated with muscle fatigue. In stroke patients, the structure of the diaphragm may shift, resulting in changes in the extremities. Pinheiro et al. reported that inspiratory muscle strength in stroke patients reached only half of that in healthy individuals, and that this reduction in inspiratory muscle function may cause functional difficulties.

In this study, ultrasonography will be used to examine the structure and function of the diaphragm and to measure muscle thickness at the end of inspiration and expiration.

All patients will be placed in the supine position, and the probe will be placed in the subcostal area between the right midclavicular line and the anterior axillary line, directed toward the head and back to reach the middle and posterior third of the diaphragm. After an optimal 2D image is obtained, the diaphragm will be evaluated and measured at end-inspiration and end-expiration. A low-frequency convex probe of 2-5 MHz will be used during the measurements.

Diaphragm contractility can be evaluated by changes in diaphragm thickness (the diaphragm thickness ratio (TR) or diaphragm thickness fraction (DTf) measured using ultrasonography).

DTf = (end-inspiration diaphragm thickness - end-expiration diaphragm thickness) / end-expiration diaphragm thickness × 100% Data Evaluation and Follow-up

Bilateral Intercostal Muscle Thickness Measurement:

Will be performed using an ultrasound device before treatment, at the 2nd week of treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).

Bilateral Diaphragm Muscle Thickness Measurement:

Will be performed using an ultrasound device before treatment, at the 2nd week of treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).

Pulmonary Function Tests:

Will be measured using spirometry before treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).

Berg Balance Scale:

Will be evaluated before treatment, at the 2nd week of treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).

Tinetti Test:

Will be evaluated before treatment, at the 2nd week of treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).

Stroke-Specific Quality of Life Scale:

Will be evaluated before treatment, at the 2nd week of treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of ischemic or hemorrhagic stroke
* Aged 18-65 years

Exclusion Criteria:

* Presence of concomitant acute or chronic lung disease
* History of thoracic or abdominal surgery
* Presence of another neuromuscular disease
* Patients with aphasia or impaired cognition
* Severe heart disease
* Active cancer
* Mini-Mental State Examination (MMSE) score ≤ 24
* Active smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years diagnosed with stroke Sample Size of the Study: 35 Stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Diaphragm muscle thickness | Will be performed using an ultrasound device before treatment, at the 2nd week of treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).
  In this study, ultrasonography will be used to examine the structure and function of the muscle and to measure muscle thickness at the end of inspiration and expiration.
Intercostal muscle thickness | Will be performed using an ultrasound device before treatment, at the 2nd week of treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).
  In this study, ultrasonography will be used to examine the structure and function of the muscle and to measure muscle thickness at the end of inspiration and expiration.

SECONDARY OUTCOMES:
Berg Balance Scale | Will be evaluated before treatment, at the 2nd week of treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).
  Berg balance scale scores range from 0 to 56. The lower your score, the more at risk you are for losing your balance. The higher your score, the better your functional mobility (ability to move effectively and safely).
Tinetti Test | Will be evaluated before treatment, at the 2nd week of treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).
  The Tinetti test has a gait score and a balance score. It uses a 3-point ordinal scale of 0, 1 and 2. Gait is scored over 12 and balance is scored over 16 totalling 28. The lower the score on the Tinetti test, the higher the risk of falling.
Stroke-Specific Quality of Life Scale | Will be evaluated before treatment, at the 2nd week of treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).
  Stroke-Specific Quality of Life Scale (SS-QoL) is used to assess the life expectancy of a stroke survivor. It is specifically designed for individuals who have had a stroke. Both personal and psychosocial effects are assessed collectively. Scores range from 49-245. Higher scores indicate better functioning.
Forced Vital Capacity | Will be measured using spirometry before treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week)
  Forced vital capacity (FVC) measures the total amount of air a person can exhale as quickly and forcefully as possible after taking a deep breath. Measured through spirometry, FVC assesses the lungs' ability to hold air and helps distinguish obstructive from restrictive lung disease.
Forced Expiratory Volume | Will be measured using spirometry before treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).
  FEV₁ (forced expiratory volume in 1 second) measures the amount of air a person can forcefully exhale in the first second after taking a deep breath. This value is used to determine the degree of airway obstruction. The FEV₁/FVC ratio is an important parameter in distinguishing obstructive and restrictive lung diseases.
Maximum Inspiratory Pressure | Will be measured using respiratory pressure meter before treatment, at the end of treatment (4th week), and 4 weeks after the completion of treatment (8th week).
  Maximum inspiratory pressure (MIP) is a measurement that evaluates the strength of the inspiratory muscles. This test measures the negative pressure created when a person breathes in at maximum effort. MIP assesses the strength of respiratory muscles, such as the diaphragm and intercostal muscles, and is used to diagnose conditions characterized by respiratory muscle weakness.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara Üniversitesi Tıp Fakültesi, Istanbul, Maltepe 34854, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No